CLINICAL TRIAL: NCT03667625
Title: The Effect of Stretching Exercises in Water and on Land on Spinal Mobility and Functional Level in Patients With Ankylosing Spondylitis
Brief Title: Stretching in Water and on Land for Patients With Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Barış Gürpınar, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DorkuzEU
Record Dates: First submitted 2018-08-27; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Ankylosing Spondylitis
Keywords: aquatherapy; stretching exercises
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aquatic group (Experimental): Aquatic multidimensional mobility exercises were given in the treatment pool at Balcova Thermal Centre, Izmir, Turkey. Group of 6-7 patients was instructed by a specialized physiotherapist twice in a week for eight weeks. The water temperature was 33-340C and the depth was between 110-140 cm, patients were asked to keep T11 level submersion during vertical exercises. Exercise span was kept 30-40 min in first 4 weeks then increased to 45-50 min with additional exercises.
  Interventions: Other: Multidimensional Mobility Exercises
- Land group (Experimental): Multidimensional mobility exercises were given at exercise unit of Dokuz Eylul University School of Physical Therapy, Izmir, Turkey. Group of 6-7 patients were instructed by a specialized physiotherapist twice in a week for eight weeks. The room temperature was 23-240C. Exercise span was kept 30-40 min in first 4 weeks then increased to 45-50 min with additional exercises.
  Interventions: Other: Multidimensional Mobility Exercises
- Control group (Active Comparator): A conventional home exercise programme was given by a specialized physiotherapist to control group. Patients were checked and encouraged to continue their programs by weekly phone calls for eight weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Multidimensional Mobility Exercises — Multidimensional mobility exercises, combined with breathing exercise protocol was established by a committee of specialized physiotherapists and rheumatologist. Land-based and aquatic-based exercises were designed according to environmental features (gravity, buoyancy, viscosity etc).
  Arms: Aquatic group; Land group
Other: Control group — A conventional home exercise programme was given by a specialized physiotherapist to control group. Patients were checked and encouraged to continue their programs by weekly phone calls for eight weeks
  Arms: Control group

SUMMARY:
The aim of the study is to investigate the effectiveness stretching exercises in ankylosing spondylitis.

DETAILED DESCRIPTION:
Ankylosing spondylitis is a chronic, progressive disease with an unknown etiology which characterize with inflammation that leads to bone fusion in spinal joints. Besides the systemic manifestations, chronic pain acquired kyphosis, diminished exercise capacity may cause pulmonary dysfunction, muscle imbalance, reduced quality of life, sleep disruptions and depression. There are strong evidence and advice on exercise should start with diagnosis. Although stretching exercises are the most common exercises in this group the literature on the effectiveness of stretching exercises is scarce. The aim of the study is to investigate the effectiveness stretching exercises in ankylosing spondylitis.

The study was carried on patients with ankylosing spondylitis followed by Division of Rheumatology and Immunology, Department of Internal Medicine, Dokuz Eylül University School of Medicine. 57 patients were assessed and randomized into two group control and intervention. Control group informed on the importance of exercise and given a home exercise brochure. The intervention group was also randomized into an aquatic and land stretching group and received stretching exercises two days a week for eight weeks. Two patients from the control group and nine patients (three from aquatic, six from land) from the intervention group were excluded.

At the end of eight weeks, except FEV1, FVC, VC all results of the intervention group improved whereas an quality of health was the only result improved in the control group. When aquatic and land stretching groups the results were improved similarly. The improvements of BASFI and MIP of the aquatic group are superior to the land group.

Home exercises are playing an important role in the management of ankylosing spondylitis. Addition of stretching exercises to home exercises enhances the effectiveness of the treatment. Aquatic stretching exercises have some benefits than land stretching exercises.

ELIGIBILITY:
Inclusion Criteria:

* AS diagnosed according to 1988 Modified New York criteria volunteered with a BASDAI score of 3 or 4

Exclusion Criteria:

* Patients followed any physical exercise within the last 3 months prior to this study, history of cardiovascular and pulmonary disease were excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09-06 (Actual)

PRIMARY OUTCOMES:
Change in Vital capacity | Baseline and 8 weeks
  Vital capacity (VC) (liter) tested with a portable spirometer (MiniSpir, Rome, Italy). The data was given as the (%) percentage of predicted value.
Change in respiratory muscle strength | Baseline and 8 weeks
  Strength of diaphragm and other inspiratory muscles was measured with maximal inspiratory pressure (MIP) (cmH2O) while strength of the abdominal muscles and other expiratory muscles was measured with maximal expiratory pressure (MEP) (cmH2O) a digital manometer (Micro RPM, Micro Medical Ltd, Kent, UK) while sitting. The data was given as the percentage (%) of predicted value.
Change in FVC | Baseline and 8 weeks
  forced vital capacity (FVC) (liter) tested with a portable spirometer (MiniSpir, Rome, Italy). The data was given as the (%) percentage of predicted value.
Change in FEV1/FVC | Baseline and 8 weeks
  forced vital capacity ratio of forced expiratory volume during the first second (FEV1/FVC), tested with a portable spirometer (MiniSpir, Rome, Italy). The data was given as the (%) percentage of predicted value.
Change in PEF | Baseline and 8 weeks
  peak expiratory flow (PEF) (liter/sec) tested with a portable spirometer (MiniSpir, Rome, Italy). The data was given as the (%) percentage of predicted value.
Change in MVV | Baseline and 8 weeks
  maximum voluntary ventilation (MVV) (liter/min) tested with a portable spirometer (MiniSpir, Rome, Italy). The data was given as the (%) percentage of predicted value.

SECONDARY OUTCOMES:
Change in functionality | Baseline and 8 weeks
  Bath ankylosing spondylitis functional index. Includes 10 questions with 10 cm visual analog scale (VAS) was used to answer the questions. The mean of the ten scales gives the BASFI score - a value between 0 and 10. The higher the BASFI score, the more severe the patient's limitation of function due to their AS
Change in disease activity | Baseline and 8 weeks
  Bath Ankylosing Spondylitis Disease Activity Index. BASDAI consists of 10 cm VAS used to answer 6 questions pertaining to the 5 major symptoms of AS: Fatigue; Spinal pain; Joint pain / swelling; Areas of localized tenderness; Morning stiffness. To give each symptom equal weighting, the mean of the two scores relating to morning stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score.The higher the BASDAI score, the more severe the patient's disability due to their AS
Change in spinal mobility | Baseline and 8 weeks
  Bath Ankylosing Spondylitis Metrology Index. Tragus to wall distance, Lumbar side flexion, Modified Schober's, Cervical rotation and Intermalleolar distance were inculuded in BASMI. The BASMI was first published in 1994 as a 2-point scale, was adapted a year later into a 10-point scale, and has more recently been proposed and validated as a linear construct. Individual scores are summed for the BASMI2 or averaged for the BASMI10 to give a final score between 0 and 10, where a higher score reflects more significant impairment of spinal mobility.
Change in muscle strength | Baseline and 8 weeks
  Upper extremity muscle strength was tested with hand dynamometer while a back and leg dynamometer was used for lower extremities and back muscle strength. Data was given kg.
Change in sleep quality | Baseline and 8 weeks
  Pittsburgh sleep quality index. It consists of nineteen questions which finally generate seven component scores: "subjective sleep quality","sleep latency", "sleep duration", "habitual sleep efficiency","sleep disturbances", "use of sleep medication" and "daytimedysfunction". These nineteen items are used for scoring. A total score above 5 is associated with a poor sleep quality
Change in depression | Baseline and 8 weeks
  Beck depression scale, a 21-item test presented in multiplechoice format, which purports to measure presence and degree of depression. Responses are made on a four-point, minimally anchored scale, ranging from 0 to 3, with 3 representing the most severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Baris GURPINAR, PhD, Principal Investigator — Dokuz Eylul University; Nursen ILCIN, PhD, Study Chair — Dokuz Eylul University; Sema SAVCI, PhD, Study Director — Dokuz Eylul University; Nurullah AKKOC, Study Director
Locations (1):
- Dokuz Eylul University School of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurpinar B, Ilcin N, Savci S, Akkoc N. Do mobility exercises in different environments have different effects in ankylosing spondylitis? Acta Reumatol Port. 2021 Oct-Dec;46(4):297-316. PMID 34962245